CLINICAL TRIAL: NCT05898152
Title: Interest of a Specific Care Pathway for the Management of Catamenial Epilepsy Catamenial Epilepsy: Status Report and Point of View of a Cohort of Patients Who for Drug-resistant Epilepsy at the TOULOUSE University Hospital
Brief Title: Interest of a Specific Care Pathway for the Management of Catamenial Epilepsy
Acronym: EPICAT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0055; 2023-A00280-45 (Other: ANSM)
Record Dates: First submitted 2023-05-15; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy Menstrual
Keywords: Catamenial epilepsy; Menstrual cycle
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with catamenial epilepsy: A questionnaire regarding the menstrual cycle and the catamenial epilepsy will be administrated to the participants.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — A collection about patient's data demographic, neurologic and gynecologic follow-up and satisfaction will be review by questionnaire. And a calendar of epileptic seizures will be completed by patients on 4 months

SUMMARY:
This is a study of patients with catamenial epilepsy. Catamenial epilepsies are defined as epileptic seizures during the menstrual cycle. Today, there are no recommendations and no care pathway for these patients. The aim of this study is to assess the number of patients reporting a link between the occurrence of their epileptic seizures and their menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients (>18 years)
* No menopausal
* Patients who have consulted in a Neurology department for refractory epilepsy
* Non opposition patient
* Affiliation to a social security scheme

Exclusion Criteria:

* Patients who understand French enough

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with catamenial epilepsy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-05-03 (Estimated); Study Completion 2024-11-03 (Estimated)

PRIMARY OUTCOMES:
Number of reporting patients | 4 months
  Number and proportion of patients reporting having a link between the onset of their epileptic seizures and their menstrual cycle based on the questionnaire they completed.

SECONDARY OUTCOMES:
Listening satisfaction | 4 months
  Questionnaire about listening satisfaction by the professional
Satisfaction of taking charge | 4 months
  Questionnaire about satisfaction of management by the professional
Rate of women with drug-resistant epilepsy | 4 months
  Collection calendar
Reconciliation of catamenial epilepsy | 4 months
  Comparison of epilepsy collection calendar and questionnaire. The questionnaire includes demographic data, neurological demographic data, their neurological and gynaecological follow-up, and also their satisfaction with their care and the information received on their pathology.
Association between catamenial epilepsy and menstrual cycle | 4 months
  Research of an association between catamenial epilepsy and menstrual cycle
Existing associations | 4 months
  Evaluate link between different factors obtained during the collection (contraceptions, epileptics, menstrual cycle disorders, etc.) and the presence of catamenial epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: Anna GOSSET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France